CLINICAL TRIAL: NCT06392282
Title: MV-140 Efficacy in Recurrent Urinary Tract Infections
Brief Title: MV-140 Efficacy in Recurrent Urinary Tract Infections in a Cohort of Portuguese Adult Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Unidade Local de Saúde Santa Maria (Other Government)
Responsible Party: Principal Investigator, Filipe Abadesso Lopes, Principal Investigator, Unidade Local de Saúde Santa Maria
Other Study IDs: 48/24
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Urinary Tract Infections
Keywords: Urinary tract infections; immunotherapy; MV-140
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: MV-140 — MV-140 use - sublingual spray approved for recurrent UTI prevention

SUMMARY:
We will access the efficacy of MV-140 immunotherapy in the prevention of recurrent urinary tract infections in a cohort of Portuguese patients.

DETAILED DESCRIPTION:
Urinary tract infections represent a highly frequent and debilitating disease, responsible for an extensive use of antibiotics for treatment and prophylaxis. Non-antibiotic therapies, such as oral vaccines, have been developed, in order to avoid antibiotic use. MV-140 is a sublingual vaccine comprised of 4 inactivated bacteria - E. coli, K. pneumoniae, E. faecalis and Proteus vulgaris. It is approved for the prevention of recurrent UTIs, with promising results in the few published results to date. The efficacy of this tool in the Portuguese population is, however, still unknown. Since the prevalence of pathogens responsible for infections and overall antibiotic use are highly variable worldwide, the results of studies conducted so far are not directly applicable in other regions. Therefore, we designed the present study which aims at assessing the efficacy of immunotherapy with MV-140 In the Portuguese population. It is a prospective observational study, in which patients will be asked to report their condition before and 1 year after therapy.

ELIGIBILITY:
Inclusion Criteria:

* At least 3 positive urine culture UTIs in the preceding 12 months
* Ability to understand and fill the informed consent

Exclusion Criteria:

I. History of genitourinary tumours II. Urinary lithiasis III. Immunodeficiency IV. Pregnancy V. Simultaneous use of any other urinary tract prevention vaccines or prophylactic antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consulted at Urology clinic with recurrent UTIs
Sampling Method: Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
UTI episodes | 1 year
  Change in number of UTI episodes

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Santa Maria, Lisbon, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: Undecided
IPD might be anonymously shared with suitable fellow researchers